CLINICAL TRIAL: NCT03318042
Title: Association Between Genotype, Polyphenol Gut Microbiota Metabotypes, and Diet in a Cohort of Children and Adolescents From the Southeast of Spain.
Brief Title: Genotype, Metabotype and Diet in a Cohort of Children and Adolescents From the Southeast of Spain.
Acronym: PolyMicroBio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: CEIP (primary school) Jara Carrillo (Alcantarilla, Murcia, Spain) (Unknown); IES (secondary school) Alcántara (Alcantarilla, Murcia, Spain) (Unknown); IMDEA Food (Other)
Responsible Party: Principal Investigator, Juan Carlos Espín de Gea, Research Professor, National Research Council, Spain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AGL2015-64124-R(1)
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Genotype, Metabotype and Dietary Habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Child-teenagers-walnuts-pomegranate (Experimental): Intake of walnuts or pomegranate juice for 3 days
  Interventions: Other: Walnuts; Other: Pomegranate juice

INTERVENTIONS:
Other: Walnuts — The group consumed a daily serving of walnuts (30 g) or 200 mL pomegranate juice for 3 days and provided a sample of urine as well as a swab specimen from the inner cheek
  Other Names: Intake of walnuts
Other: Pomegranate juice — Those volunteers who were allergic to nuts consumed 200 mL pomegranate juice daily for 3 days and provided a sample of urine as well as a swab specimen from the inner cheek
  Other Names: Intake of pomegranate juice

SUMMARY:
The objective of this study is to investigate the possible association between 60 SNPs related to obesity, metabolism and cardiovascular disease with BMI, intestinal microbiota and adherence to the Mediterranean diet in a cohort of children and adolescents from the southeast of Spain.

DETAILED DESCRIPTION:
The objective of this study is to investigate the possible association between 60 single nucleotide polymorphisms (SNPs) related to obesity, metabolism and cardiovascular disease with the body mass index (BMI), intestinal microbiota related to the metabolism of polyphehnos and adherence to the Mediterranean diet in a cohort of children and adolescents from the southeast of Spain.

The volunteers (n=423) with ages ranging from 5 to 18 years consumed for three days a daily serving of walnuts (30g) and provided a sample of urine (to determine mirobial-derived metabolites from walnut polyphenols) as well as a swab specimen from the inner cheek to provide DNA for further genotyping.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 5 to 18 years.
* Informed consent signed by the parent / legal representative, and by volunteers who are already 18 years old.

Exclusion Criteria:

* Known or suspected allergy or intolerance to nuts or pomegranate.
* Intake of antibiotics 1 month before the start of the study.
* If the participant could perceive stress or psychological damage due to his participation.
* Any other circumstance different from previous ones (illness, etc.), according to which it is considered that the intervention in the study may involve some type of affectation.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 423 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-11-02 (Actual)

PRIMARY OUTCOMES:
Polyphenol metabotypes | 1 to 3 months
  Type of ellagic acid-derived microbial metabolites in urine

SECONDARY OUTCOMES:
Genotype | 1 to 6 months
  Detection of 60 SNPs related to obesity, metabolism and cardiovascular disease
Adherence to Mediterranean diet | 1 to 3 months
  Evaluation of the adherence to Mediterranean diet using validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Juan C. Espin, PhD, Principal Investigator — Spanish National Research Council (CSIC)
Locations (1):
- Cebas-Csic, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No